CLINICAL TRIAL: NCT02076477
Title: The Prospective,Multicenter,Randomized Controlled Clinical Study of the Optimal Intervention Time of Radiotherapy for Oligometastatic Stage IV Non-small Cell Lung Cancer（NSCLC）
Brief Title: The Optimal Intervention Time of Radiotherapy for Oligometastatic Stage IV Non-small Cell Lung Cancer（NSCLC）
Acronym: OITROLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Mianyang Central Hospital (Other); Cancer Hospital of Guizhou Province (Other)
Responsible Party: Principal Investigator, LI TAO, Section Head, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: scch201402
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Oligo-metastatic Stage IV Non-small Cell Lung Cancer
Keywords: intervention time; radiotherapy; oligometastatic; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy; Docetaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients receive concurrent chemoradiotherapy at first。Patients also receive chemotherapy every 3-4 weeks for two cycles after concurrent chemoradiotherapy.
  chemotherapy：（1） squamous cell carcinoma：Docetaxel 60mg/m2 d1+Cisplatin 25mg/m2 d1-3.（2）non squamous cell carcinoma： pemetrexed 500mg/m2 d1+Cisplatin 25mg/m2 d1-3.
  Interventions: Radiation: concurrent chemoradiotherapy; Drug: Docetaxel; Drug: pemetrexed; Drug: Cisplatin
- Arm B (Active Comparator): Patients receive neoadjuvant chemotherapy every 3-4 weeks for two cycles at first.Patients then receive concurrent chemoradiotherapy after neoadjuvant chemotherapy.
  chemotherapy：（1） squamous cell carcinoma：Docetaxel 60mg/m2 d1+Cisplatin 25mg/m2 d1-3.（2）non squamous cell carcinoma： pemetrexed 500mg/m2 d1+Cisplatin 25mg/m2 d1-3.
  Interventions: Radiation: concurrent chemoradiotherapy; Drug: Docetaxel; Drug: pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Radiation: concurrent chemoradiotherapy — Radiation（image-guided radiotherapy）：（1）primary tumors≤3cm，Hypofractionated radiation therapy，accumulated dose BED ≥80Gy （central lung cancer），BED ≥100Gy（Peripheral lung cancer）.（2）primary tumors>3cm，conventional fractionated radiotherapy，accumulated dose BED=60-66Gy/30-33f.（3） regional lymph node:conventional fractionated radiotherapy，accumulated dose BED=60-66Gy/30-33f.（4） Brain metastases： whole brain radiation therapy，36Gy/12f,Intracranial metastases，48Gy/12f.（5） bone metastasis：36 Gy/12f.
Drug: Docetaxel — Docetaxel:60mg/m2 d1,Given IV
Drug: pemetrexed — pemetrexed: 500mg/m2 d1,Given IV
Drug: Cisplatin — Cisplatin：25mg/m2 d1-3，Given IV

SUMMARY:
This study evaluates the optimal intervention time of radiotherapy for oligometastatic stage iv lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old , male or female
* Pathologically or cytologically proven oligometastatic stage IV NSCLC non-small cell lung cancer（NSCLC）
* Primary tumors can be measured
* Distant organ metastases number ≤ 5
* Karnofsky score >70,Zubrod performance status 0-1
* Estimated life expectancy of at least 12 weeks
* reproductive age women should ensure that before entering the study period contraception
* Hemoglobin≥10.0g/dL,WBC≥ 4000 cells/mm³,Platelet count≥100,000 cells/mm³
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal,bilirubin normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Patients have good compliance to treatment and follow-up of acceptance.

Exclusion Criteria:

* Allergic to pemetrexed, cisplatin, docetaxel and contrast medium
* Distant metastases organs > 5
* The primary tumor or lymph node already received surgical treatment (except for biopsy)
* Patient who received radiotherapy for primary tumor or lymph node
* Patient who received the the epidermal growth factor targeted therapy
* Patient who received chemotherapy or immunotherapy
* Patient who suffered from other malignant tumor
* Patient who have taken other drug test within 1 month
* Pregnant woman or Lactating Women and Women in productive age who refuse to take contraception in observation period
* Subject with a severe allergic history or idiosyncratic
* Subject with severe pulmonary and cardiopathic disease history
* Refuse or incapable to sign the informed consent form of participating this trial
* Drug abuse or alcohol addicted
* Subject with a Personality or psychiatric diseases, people with no legal capacity or people with limited capacity for civil conduct

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
short-term effects（The response rate，RR） | 3 months after the end of the treatment
  Response Evaluation Criteria In Solid Tumors (RECIST)

SECONDARY OUTCOMES:
PFS（progression-free survival） | up to 3 years
Quality of life (QOL) | up to 3 years
  Quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Trial Outcome Index (FACT-TOI) and lung cancer subscale (LCS)
esophagitis and pneumonitis | up to 3 years
  Grade 3-5 esophagitis and pneumonitis adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0
Other grade 3-5 adverse events | up to 3 years
  Other grade 3-5 adverse events as assessed by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: JIAHUA LV, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute; XIAOHU WANG, MD, PhD, Principal Investigator — Gansu Cancer Hospital; XIAOBO DU, MD, PhD, Principal Investigator — Mianyang Central Hospital; BING LU, MD.PhD, Principal Investigator — Cancer Hospital of Guizhou Province
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China